CLINICAL TRIAL: NCT01813305
Title: A Randomized,Double-Blind,Vehicle-controlled,Parallel,Phase II Study to Evaluate Efficacy and Safety of CSTC1 in Patient With Diabetic Foot Ulcers
Brief Title: CSTC1 for Diabetic Foot Ulcers Phase II Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Charsire Biotechnology Corp. (Industry)
Collaborators: ASKLEP Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CSTC1-01
Record Dates: First submitted 2013-03-12; First posted 2013-03-18 (Estimated); Results first posted 2022-04-12 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-02

CONDITIONS: Diabetic Foot Ulcer; Diabetes Mellitus; Wounds
Keywords: Diabetic Foot Ulcer; Diabetes Mellitus; Debridement; Standard of Care; wounds
MeSH Terms: conditions — Diabetic Foot; Diabetes Mellitus; Wounds and Injuries

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- CSTC1 (Active Comparator): CSTC1 (vapor fraction from seeds of Glycine max (L.) Merr. and composition thereof), topical, two times daily
  Interventions: Drug: CSTC1
- CSTC1 Matched vehicle (Placebo Comparator): Matched vehicle, topical, two times daily
  Interventions: Drug: CSTC1 Matched vehicle

INTERVENTIONS:
Drug: CSTC1 — vapor fraction from seeds of Glycine max (L.) Merr. and composition thereof
  Arms: CSTC1
Drug: CSTC1 Matched vehicle
  Arms: CSTC1 Matched vehicle

SUMMARY:
The objective of this study is to evaluate the efficacy and safety of CSTC1 in patient with diabetic foot ulcers.

DETAILED DESCRIPTION:
This study was designed as a randomized, double-blind, vehicle-controlled, multiple-center, and parallel trial to evaluate the efficacy and safety of CSTC1 in patients with diabetic foot ulcers (DFU). In each study site, eligible patients were randomized in a 4:1 ratio to receive either one of the topical applications of CSTC1 or CSTC1 matched vehicle, topical application on target diabetic foot ulcer (DFU), 2 times daily.

The treatment duration for each subject was 12 weeks or up to confirmed complete ulcer closure, whichever comes first. That was, subjects would receive treatment for at most 12 weeks, which consists of 8 visits located at weeks 1, 2, 3, 4, 6, 8, 10, and 12. Subjects who achieved confirmed complete ulcer closure during the treatment period would be arranged for a 12 week post-treatment follow-up. Subjects failed to achieve complete ulcer closure at week-12 visit would be arranged for 4 weeks of safety follow-up. If confirmation of complete ulcer closure was reached at a week-14 visit, the subject would continue the post-treatment follow-up visit until week-24 visit. Otherwise, the subject would be arranged for safety follow-up until week-16 visit.

ELIGIBILITY:
Inclusion Criteria:

* With either gender aged at least 20 years old;
* With a diabetic ulcer (which is defined as the target ulcer) on the foot and not healing for at least 2 weeks;
* The target ulcer is classified as grade 1 or 2 ulcer according to modified Wagner system;
* The target ulcer should show "infection control" at investigator's discretion;
* Subject should be free of any necrosis or infection in soft and bone tissue;
* Subject has signed the written informed consent form

Exclusion Criteria:

* With active osteomyelitis;
* With target ulcer size decreased by at least 50% after at least 2 weeks of standard-of-care-only period or any other recorded regular therapy before Randomization visit;
* With poor nutritional status (albumin < 3g/dl), poor diabetic control (HbA1c > 12%), anemia (hemoglobin<10 g/dL), a leukocyte counts < 1,000/mm3, abnormal liver function (AST, ALT>3 x upper limit of normal range);
* Requiring treatment with corticosteroids, immunosuppressive or chemotherapeutic agents;
* Presence of necrosis, purulence or sinus tracts that cannot be removed by debridement;
* Receiving revascularization surgery performed <8 weeks before entry in the study;
* With known or suspected hypersensitivity to any ingredients of study product and vehicle;
* With coronary heart disease with myocardial infarction, coronary artery bypass graft (CABG), or percutaneous transluminal coronary angioplasty (PTCA) within 3 months prior to study;
* Pregnant or lactating or premenopausal with childbearing potential but not taking reliable contraceptive method(s) during the study period;
* Enrollment in any investigational drug trial within 4 weeks before entering this study;
* With any uncontrolled illness judged by the investigator that entering the trial may be detrimental to the subject.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2014-07-09 (Actual); Primary Completion 2020-01-07 (Actual); Study Completion 2020-01-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Su-Shin Lee, MD, Principal Investigator — Kaohsiung Medical University Chung-Ho Memorial Hospital
Locations (1):
- Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The planned sample size was determined to be 80 versus 20 subjects (4:1 ratio) for treatment versus vehicle groups, 100 subjects in total. To ensure the completion of 100 evaluable subjects, around 125 subjects were planned to be recruited. In the actual trial, a total of 137 subjects were screened, with 124 meeting the criteria followed by randomization to CSTC1 group (n = 98) or Vehicle group (n = 26).
Period: Overall Study
Arm/Group | CSTC1 | CSTC1 Matched Vehicle
Started | 98 | 26
Completed | 63 | 18
Not Completed | 35 | 8
Not completed — Withdrawal by Subject | 12 | 5
Not completed — Safety Concern | 4 | 0
Not completed — Ulcer became worse | 4 | 0
Not completed — Physician Decision | 4 | 0
Not completed — Lost to Follow-up | 3 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Prohibited Medication Administration or Condition Worsening | 7 | 2

BASELINE CHARACTERISTICS:
Population: The baseline analysis population was based on ITT population.
Groups:
- Total: Total of all reporting groups
Arm/Group | CSTC1 | CSTC1 Matched Vehicle | Total
Number analyzed (Participants) | 98 | 26 | 124
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.1 (13.79) | 58.6 (11.84) | 58.2 (13.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 17 | 84
  Male | 31 | 9 | 40
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Taiwan | 98 | 26 | 124
Baseline Diabetic Foot Target Ulcer Size [Count of Participants; unit: Participants]
  > 1 ~ 1.5 cm^2 | 27 | 5 | 32
  > 1.5 ~ 2 cm^2 | 11 | 4 | 15
  > 2 ~ 3 cm^2 | 15 | 4 | 19
  > 3 ~ 4 cm^2 | 14 | 2 | 16
  > 4 ~ 5 cm^2 | 8 | 4 | 12
  > 5 ~ 10 cm^2 | 15 | 4 | 19
  > 10 ~ 15 cm^2 | 4 | 1 | 5
  > 15 ~ 20 cm^2 | 2 | 1 | 3
  > 20 cm^2 | 2 | 1 | 3
Maximum Grade of Foot Ulcers [Count of Participants; unit: Participants] — The target ulcer is classified as Grade 0 ~ 5 according to modified Wagner system. The Wagner system assesses ulcer depth and the presence of osteomyelitis or gangrene by using the following grades: grade 0 (pre-or postulcerative lesion), grade 1 (partial/full thickness ulcer), grade 2 (probing to tendon or capsule), grade 3 (deep with osteitis), grade 4 (partial foot gangrene), and grade 5 (whole foot gangrene). Higher grades were considered worse.
  Participants
    Grade 1 | 15 | 4 | 19
    Grade 2 | 83 | 22 | 105
Baseline Target Ulcer Size [Mean (Standard Deviation); unit: cm^2] | 4.37 (5.471) | 5.15 (5.531) | 4.53 (5.470)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Complete Ulcer Closure During the Treatment Period
Description: Complete ulcer closure is defined as 100% skin re-epithelialization without drainage or dressing requirements confirmed at the coming visits 2 weeks apart. The treatment period is until 12 weeks or up to confirmation of complete ulcer closure. Subjects with complete ulcer closure at Week 12 and confirmed at Week 14 were considered as success.
Time Frame: Baseline to 14 weeks
Population: All randomized subjects who have received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | CSTC1 | CSTC1 Matched Vehicle
Number analyzed (Participants) | 98 | 26
Participants | 32 | 4

2. Secondary Outcome: The Ulcer Closure Time
Description: Defined as the time to complete ulcer closure.
Time Frame: 24 weeks
Population: All randomized subjects who have received at least one dose of study medication.
Measure: Mean (Standard Error); unit: Days
Arm/Group | CSTC1 | CSTC1 Matched Vehicle
Number analyzed (Participants) | 98 | 26
Days | 87 (2.2) | 92 (3.2)

3. Secondary Outcome: The Accumulated Participant Counts With Complete Ulcer Closure
Description: Complete ulcer closure is defined as 100% skin re-epithelialization without drainage or dressing requirements observed for at the last two consecutive study visits 2 weeks apart. The count of participants with complete ulcer closure at each post-treatment visit is provided.
Time Frame: 24 weeks
Population: All randomized patients who have received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | CSTC1 | CSTC1 Matched Vehicle
Number analyzed (Participants) | 98 | 26
Participants
  Week 1 | 0 | 0
  Week 2 | 0 | 0
  Week 3 | 0 | 0
  Week 4 | 0 | 0
  Week 6 | 2 | 1
  Week 8 | 9 | 1
  Week 10 | 13 | 1
  Week 12 | 22 | 2
  Week 14 | 32 | 4
  Week 16 | 35 | 7
  Week 20 | 35 | 7
  Week 24 | 36 | 6

4. Secondary Outcome: Percentage Change in Ulcer Size for Each Post-treatment Visit
Description: The proportion of ulcer closure is calculated as (Ulcer size at post-treatment visit - Ulcer size at baseline)/(Ulcer size at baseline). This proportion was then multiplied by 100 to calculate the percentage change in ulcer size for each post-treatment visit. The percentage change in ulcer size for each post-treatment visit are presented.
Time Frame: baseline and 24 weeks
Population: All randomized patients who have received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | CSTC1 | CSTC1 Matched Vehicle
Number analyzed (Participants) | 98 | 26
percent change
  Week 1 | -15.2 (28.31) | -16.3 (25.09)
  Week 2 | -28.3 (30.32) | -21.7 (32.82)
  Week 3 | -36.3 (34.93) | -29.1 (41.00)
  Week 4 | -46.6 (35.15) | -32.8 (36.90)
  Week 6 | -53.6 (40.13) | -44.8 (41.11)
  Week 8 | -56.7 (49.96) | -47.0 (46.67)
  Week 10 | -61.7 (47.01) | -51.8 (44.85)
  Week 12 | -66.3 (41.91) | -54.2 (56.52)
  Week 14 | -69.1 (39.09) | -57.6 (57.54)
  Week 16 | -69.8 (38.40) | -59.1 (60.05)
  Week 20 | -70.4 (38.60) | -59.1 (60.05)
  Week 24 | -70.2 (38.52) | -59.0 (59.95)

5. Other Pre Specified Outcome: Number of Participants With Adverse Events
Description: An AE is any untoward medical occurrence in a patient or clinical investigation participant administered a study medication and that does not necessarily have a causal relationship with this treatment. An AE can, therefore, be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of study medication, whether or not related to the study medication. AE data was collected from Screening visit to Final visit (up to 24 weeks).
Time Frame: 24 weeks
Population: All randomized patients who have received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | CSTC1 | CSTC1 Matched Vehicle
Number analyzed (Participants) | 98 | 26
Participants | 80 | 22

6. Other Pre Specified Outcome: Number of Participants With Physical Abnormality Finding at the Visits
Description: Physical examinations in this study included the following items: general appearance, skin, eyes, ears, nose, throat, head and neck, heart, joints, chest and lungs, abdomen, lymph nodes, musculoskeletal, nervous system, and others. Physical examinations were conducted from Screening visit to Final visit (up to 24 weeks). If at least one of physical examinations was identified in the subject, the subject was included in physical abnormalities calculation.
Time Frame: 24 weeks
Population: All randomized patients who have received at least one dose study medication.
Measure: Number; unit: participants
Arm/Group | CSTC1 | CSTC1 Matched Vehicle
Number analyzed (Participants) | 98 | 26
participants
  Baseline (Day 1) | 57 | 18
  Week 1 | 57 | 18
  Week 2: number analyzed (Participants) | 95 | 26
  Week 2 | 57 | 18
  Week 3: number analyzed (Participants) | 94 | 24
  Week 3 | 59 | 16
  Week 4: number analyzed (Participants) | 93 | 24
  Week 4 | 57 | 16
  Week 6: number analyzed (Participants) | 91 | 25
  Week 6 | 57 | 17
  Week 8: number analyzed (Participants) | 86 | 21
  Week 8 | 52 | 16
  Week 10: number analyzed (Participants) | 74 | 21
  Week 10 | 45 | 16
  Week 12: number analyzed (Participants) | 67 | 21
  Week 12 | 41 | 16
  Week 14: number analyzed (Participants) | 69 | 18
  Week 14 | 43 | 12
  Week 16: number analyzed (Participants) | 68 | 18
  Week 16 | 42 | 12
  Week 20: number analyzed (Participants) | 30 | 4
  Week 20 | 18 | 2
  Week 24: number analyzed (Participants) | 27 | 4
  Week 24 | 15 | 2

7. Other Pre Specified Outcome: Number of Participants With Relieved, Unchanged, or Worsen Values in Laboratory Test at Week 12 Compared to Baseline
Description: Laboratory examination to be measured in this study consisted of hematology (hemoglobin, hematocrit, RBC, platelet, WBC with differential counts) and biochemistry (Aspartate Transaminase (AST), Alanine Transaminase (ALT), fasting glucose, HbA1c, serum creatinine, blood urea nitrogen (BUN), albumin). The laboratory examinations were conducted at the Screening visit, baseline, and Week 12. Patients' laboratory change from baseline to Week 12 was documented as relieved, unchanged, worsened (MH), or worsened (AE). The "worsened" means that the laboratory values were normal or non clinically significant (NCS) at baseline but change to clinically significant at Week 12. If the worsen situation was found, the clinically significant worsening changes were classified as related to medical history (MH) or adverse events (AE).
Time Frame: baseline and 12 weeks
Population: All randomized patients who have received at least one dose study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | CSTC1 | CSTC1 Matched Vehicle
Number analyzed (Participants) | 98 | 26
Participants
  White blood cells (10^9/L): number analyzed (Participants) | 88 | 22
  White blood cells (10^9/L): Relieved | 0 | 0
  White blood cells (10^9/L): Unchanged | 81 | 22
  White blood cells (10^9/L): Worsened (MH) | 2 | 0
  White blood cells (10^9/L): Worsened (AE) | 5 | 0
  Neutrophils (%): number analyzed (Participants) | 87 | 22
  Neutrophils (%): Relieved | 0 | 0
  Neutrophils (%): Unchanged | 84 | 22
  Neutrophils (%): Worsened (MH) | 2 | 0
  Neutrophils (%): Worsened (AE) | 1 | 0
  Eosinophils (%): number analyzed (Participants) | 87 | 22
  Eosinophils (%): Relieved | 0 | 0
  Eosinophils (%): Unchanged | 87 | 22
  Eosinophils (%): Worsened (MH) | 0 | 0
  Eosinophils (%): Worsened (AE) | 0 | 0
  Basophils (%): number analyzed (Participants) | 87 | 22
  Basophils (%): Relieved | 0 | 0
  Basophils (%): Unchanged | 87 | 22
  Basophils (%): Worsened (MH) | 0 | 0
  Basophils (%): Worsened (AE) | 0 | 0
  Lymphocytes (%): number analyzed (Participants) | 87 | 22
  Lymphocytes (%): Relieved | 0 | 0
  Lymphocytes (%): Unchanged | 83 | 22
  Lymphocytes (%): Worsened (MH) | 2 | 0
  Lymphocytes (%): Worsened (AE) | 2 | 0
  Monocytes (%): number analyzed (Participants) | 87 | 22
  Monocytes (%): Relieved | 0 | 0
  Monocytes (%): Unchanged | 87 | 22
  Monocytes (%): Worsened (MH) | 0 | 0
  Monocytes (%): Worsened (AE) | 0 | 0
  Red Blood Cells (^12/L): number analyzed (Participants) | 88 | 22
  Red Blood Cells (^12/L): Relieved | 2 | 0
  Red Blood Cells (^12/L): Unchanged | 81 | 21
  Red Blood Cells (^12/L): Worsened (MH) | 5 | 1
  Red Blood Cells (^12/L): Worsened (AE) | 0 | 0
  Hemoglobin (g/mL): number analyzed (Participants) | 88 | 22
  Hemoglobin (g/mL): Relieved | 3 | 0
  Hemoglobin (g/mL): Unchanged | 80 | 21
  Hemoglobin (g/mL): Worsened (MH) | 5 | 1
  Hemoglobin (g/mL): Worsened (AE) | 0 | 0
  Hematocrit (%): number analyzed (Participants) | 88 | 22
  Hematocrit (%): Relieved | 2 | 0
  Hematocrit (%): Unchanged | 82 | 21
  Hematocrit (%): Worsened (MH) | 4 | 1
  Hematocrit (%): Worsened (AE) | 0 | 0
  Platelets (10^9/L): number analyzed (Participants) | 88 | 22
  Platelets (10^9/L): Relieved | 0 | 0
  Platelets (10^9/L): Unchanged | 86 | 22
  Platelets (10^9/L): Worsened (MH) | 2 | 0
  Platelets (10^9/L): Worsened (AE) | 0 | 0
  Hemoglobin A1C (%): number analyzed (Participants) | 88 | 22
  Hemoglobin A1C (%): Relieved | 5 | 0
  Hemoglobin A1C (%): Unchanged | 79 | 21
  Hemoglobin A1C (%): Worsened (MH) | 4 | 1
  Hemoglobin A1C (%): Worsened (AE) | 0 | 0
  Aspartate Aminotransferase (U/L): number analyzed (Participants) | 87 | 22
  Aspartate Aminotransferase (U/L): Relieved | 1 | 0
  Aspartate Aminotransferase (U/L): Unchanged | 85 | 22
  Aspartate Aminotransferase (U/L): Worsened (MH) | 1 | 0
  Aspartate Aminotransferase (U/L): Worsened (AE) | 0 | 0
  Alanine Aminotransferase (U/L): number analyzed (Participants) | 88 | 22
  Alanine Aminotransferase (U/L): Relieved | 1 | 0
  Alanine Aminotransferase (U/L): Unchanged | 86 | 22
  Alanine Aminotransferase (U/L): Worsened (MH) | 1 | 0
  Alanine Aminotransferase (U/L): Worsened (AE) | 0 | 0
  Blood Urea Nitrogen (U/L): number analyzed (Participants) | 88 | 22
  Blood Urea Nitrogen (U/L): Relieved | 6 | 2
  Blood Urea Nitrogen (U/L): Unchanged | 77 | 19
  Blood Urea Nitrogen (U/L): Worsened (MH) | 5 | 1
  Blood Urea Nitrogen (U/L): Worsened (AE) | 0 | 0
  Creatinine (umol/L): number analyzed (Participants) | 88 | 22
  Creatinine (umol/L): Relieved | 6 | 1
  Creatinine (umol/L): Unchanged | 78 | 21
  Creatinine (umol/L): Worsened (MH) | 4 | 0
  Creatinine (umol/L): Worsened (AE) | 0 | 0
  Glucose (mg/dL): number analyzed (Participants) | 88 | 22
  Glucose (mg/dL): Relieved | 13 | 1
  Glucose (mg/dL): Unchanged | 66 | 18
  Glucose (mg/dL): Worsened (MH) | 9 | 3
  Glucose (mg/dL): Worsened (AE) | 0 | 0

8. Other Pre Specified Outcome: Blood Pressure Change From Baseline to Week 24
Description: Vital signs measurement consisted of blood pressures, pulse rate, respiratory rate, and body temperature. Among them, blood pressure (systolic/diastolic) were obtained after the subject has been at rest for at least 5 minutes in a sitting position. The vital sign data was collected from Screening visit to Final visit (up to 24 weeks). The mean changes of Final visit to baseline in vital signs were presented (value at 24 weeks minus value at baseline).
Time Frame: baseline and 24 weeks
Population: All randomized patients who have received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | CSTC1 | CSTC1 Matched Vehicle
Number analyzed (Participants) | 98 | 26
mmHg
  Systolic Blood Pressure [mmHg]: number analyzed (Participants) | 27 | 4
  Systolic Blood Pressure [mmHg] | -3.67 (27.088) | -20.00 (34.137)
  Diastolic Blood Pressure [mmHg]: number analyzed (Participants) | 27 | 4
  Diastolic Blood Pressure [mmHg] | 1.41 (13.882) | -6.25 (4.646)

9. Other Pre Specified Outcome: Pulse Rate Change From Baseline to Week 24
Description: Vital signs measurement consisted of blood pressures, pulse rate, respiratory rate, and body temperature. Among them, pulse rates were obtained after the subject has been at rest for at least 5 minutes in a sitting position. The vital sign data was collected from Screening visit to Final visit (up to 24 weeks). The mean changes of Final visit to baseline in vital signs were presented (value at 24 weeks minus value at baseline).
Time Frame: baseline and 24 weeks
Population: All randomized patients who have received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: beats/min
Groups:
- CSTC1 Matched Vehicle: Matched vehicle, topical, two times daily
  CSTC1 Matched vehicle
Arm/Group | CSTC1 | CSTC1 Matched Vehicle
Number analyzed (Participants) | 27 | 4
beats/min | 4.00 (9.899) | -1.25 (9.323)

10. Other Pre Specified Outcome: Body Temperature Change From Baseline to Week 24
Description: Vital signs measurement consisted of blood pressures, pulse rate, respiratory rate, and body temperature. Among them, body temperature were obtained after the subject has been at rest for at least 5 minutes in a sitting position. The vital sign data was collected from Screening visit to Final visit (up to 24 weeks). The mean changes of Final visit to baseline in vital signs were presented (value at 24 weeks minus value at baseline).
Time Frame: baseline and 24 weeks
Population: All randomized patients who have received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: degrees Celsius
Arm/Group | CSTC1 | CSTC1 Matched Vehicle
Number analyzed (Participants) | 27 | 4
degrees Celsius | 0.08 (0.468) | 0.33 (0.377)

11. Other Pre Specified Outcome: Respiratory Rate Change From Baseline to Week 24
Description: Vital signs measurement consisted of blood pressures, pulse rate, respiratory rate, and body temperature. Among them, respiratory rate were obtained after the subject has been at rest for at least 5 minutes in a sitting position. The vital sign data was collected from Screening visit to Final visit (up to 24 weeks). The mean changes of Final visit to baseline in vital signs were presented (value at 24 weeks minus value at baseline).
Time Frame: baseline and 24 weeks
Population: All randomized patients who have received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: breaths/min
Arm/Group | CSTC1 | CSTC1 Matched Vehicle
Number analyzed (Participants) | 27 | 4
breaths/min | -0.11 (1.672) | -3.25 (3.862)

12. Post Hoc Outcome: Time to Achieve ≥ 50% Reduction in Target Ulcer Size
Description: The proportion of ulcer closure is calculated as (Ulcer size at post-treatment visit - Ulcer size at baseline)/(Ulcer size at baseline). Time to achieve ≥ 50% reduction in target ulcer size was measured from Screening visit to Final visit (up to 24 weeks).
Time Frame: 24 weeks
Population: All randomized patients who have received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | CSTC1 | CSTC1 Matched Vehicle
Number analyzed (Participants) | 98 | 26
Days | 42 (3.3) | 52 (7.1)

13. Post Hoc Outcome: The Response Rate of the Target Ulcer Size Reduction ≥ 50%
Description: The proportion of ulcer closure is calculated as (Ulcer size at post-treatment visit - Ulcer size at baseline)/(Ulcer size at baseline). A subject who had target ulcer closure ≥ 50% was counted as a responder. The non-responders included subjects whose target ulcer closure size less than 50% before 12 weeks.
Time Frame: 12 weeks
Population: All randomized patients who have received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | CSTC1 | CSTC1 Matched Vehicle
Number analyzed (Participants) | 98 | 26
Participants
  Responder | 77 | 18
  Non-Responder | 21 | 8

14. Post Hoc Outcome: Time to Achieve ≥90% Reduction in Target Ulcer Size
Description: The proportion of ulcer closure is calculated as (Ulcer size at post-treatment visit - Ulcer size at baseline)/(Ulcer size at baseline). Time to achieve ≥ 90% reduction in target ulcer size was analyzed in the subjects.
Time Frame: 24 weeks
Population: All randomized patients who have received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | CSTC1 | CSTC1 Matched Vehicle
Number analyzed (Participants) | 98 | 26
Days | 73 (2.9) | 84 (4.4)

15. Post Hoc Outcome: The Response Rate of the Target Ulcer Size Reduction ≥ 90%
Description: Subjects with ulcer closure size ≥ 90% compared to the baseline at a Week 12 were considered as a responder. A subject whose target ulcer size reduction was less than 90% was counted as a non-responder. The percentage of repsonders and non-responders were presented.
Time Frame: 12 weeks
Population: All randomized patients who have received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | CSTC1 | CSTC1 Matched Vehicle
Number analyzed (Participants) | 98 | 26
Participants
  Responder | 49 | 12
  Non-Responder | 49 | 14

ADVERSE EVENTS:
Time Frame: AE data was collected from Screening visit to Final visit (up to 24 weeks)
Description: All enrolled subjects were used for the analysis of AE and SAE
Arm/Group | CSTC1 | CSTC1 Matched Vehicle
All-Cause Mortality (participants affected / at risk) | 2/98 | 1/26
Serious Adverse Events (participants affected / at risk) | 20/98 | 3/26
Other Adverse Events (participants affected / at risk) | 44/98 | 13/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CSTC1 (N=98) | CSTC1 Matched Vehicle (N=26)
Cellulitis (Infections and infestations) | 5 (5) | 1 (1)
Abdominal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Wound sepsis (Infections and infestations) | 1 (1) | 0 (0)
Diabetic gangrene (Infections and infestations) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Orthostatic hypotension (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 1 (1) | 0 (0)
Application site cellulitis (Infections and infestations) | 2 (2) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 1 (1)
Impaired healing (General disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Streptococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CSTC1 (N=98) | CSTC1 Matched Vehicle (N=26)
Cataract (Eye disorders) | 5 (5) | 0 (0)
Application site erosion (General disorders) | 6 (7) | 0 (0)
Peripheral swelling (General disorders) | 4 (4) | 2 (2)
Nasopharyngitis (Infections and infestations) | 7 (7) | 2 (2)
Limb injury (Injury, poisoning and procedural complications) | 17 (31) | 7 (12)
Skin abrasion (Injury, poisoning and procedural complications) | 5 (5) | 1 (1)
Wound complication (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Skin wound (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-23): https://cdn.clinicaltrials.gov/large-docs/05/NCT01813305/Prot_SAP_000.pdf